CLINICAL TRIAL: NCT02507700
Title: Popliteal Block for Postoperative Pain in Knee-ankle Soft Tissue Surgery in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Associate Professor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DiskapiTRH 2015
Record Dates: First submitted 2015-07-15; First posted 2015-07-24 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Postoperative Pain; Cerebral Palsy
Keywords: nerve block
MeSH Terms: conditions — Pain, Postoperative; Cerebral Palsy | interventions — Sevoflurane; Ultrasonography; Bupivacaine; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- popliteal block (Active Comparator): Popliteal block will be performed with a single dose of 0.3 ml·kg(-1) of 0.25% bupivacaine.
  Interventions: Procedure: Popliteal block; Drug: Sevoflurane; Device: Ultrasound; Drug: bupivacaine; Other: Laryngeal mask airway
- Plaster cover (Sham Comparator): Only plaster cover will be applied without nerve block for sham procedure.
  Interventions: Drug: Sevoflurane; Other: Plaster cover; Other: Laryngeal mask airway

INTERVENTIONS:
Procedure: Popliteal block — In group P, popliteal block will be performed with ultrasound guidence.
  Arms: popliteal block
Drug: Sevoflurane — Sevoflurane will be used to all patient's for anesthesia induction and maintenance
Device: Ultrasound — For recognize the nerve (sciatic nerve), ultrasound will be used in group P.
  Arms: popliteal block
Other: Plaster cover — Plaster cover will be used to control group for sham procedure
  Arms: Plaster cover
Drug: bupivacaine — Bupivacaine 0.25% will be performed for popliteal block to group P.
  Arms: popliteal block
Other: Laryngeal mask airway — After anesthesia induction, laryngeal mask airway will be inserted to all patients

SUMMARY:
Popliteal block is a technique for providing postoperative pain management in children. In this randomized double-blinded study, the investigators evaluated the effects of preoperative popliteal nerve block on postoperative pain and analgesic requirement in children with cerebral palsy (CP) undergoing knee-anckle soft tissue surgery. The Wong Baker faces scale and skin conductance fluctuations will be assessed.

DETAILED DESCRIPTION:
Sevoflurane will be used for anesthesia induction and maintance. Laryngeal mask airway will be placed without neuromuscular blocking agent. In group P (popliteal block), a single dose of 0.3ml.kg(-1) of 0.25% bupivacaine will be performed for popiteal nerve block (with ultrasound guidence). In group C ( control), only plaster cover will be applied without nerve block for sham procedure to provide double-blinded study. Intraoperative heart rate, mean arterial pressure, BIS (bispectral index) values, sevoflurane consumption will be recorded ten minutes interval. Wong Baker faces scale and skin conductance fluctuations will be recorded at postoperative 0, 10th min, 20th min , 1st h, 4th h, 12th h qnd 24th h. Total analgesic consumption (paracetamol orally ) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Scheduled for knee and ankle surgery

Exclusion Criteria:

* Autonomic neuropathy
* Medication with anticholinergic drugs
* Continuous infusion of vasoactive drugs

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment via Wong Baker faces scale | The patients will be followed up to 24 hours
The number of fluctuations of skin conductance per second (NFSC). | The patients will be followed up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Taylan Akkaya, Study Chair — Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital; Mesut Bakır, Study Chair — Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Ledowski T, Bromilow J, Wu J, Paech MJ, Storm H, Schug SA. The assessment of postoperative pain by monitoring skin conductance: results of a prospective study. Anaesthesia. 2007 Oct;62(10):989-93. doi: 10.1111/j.1365-2044.2007.05191.x. PMID 17845649
- [Result] Johnston BM, Gunn TR, Gluckman PD. Surface cooling rapidly induces coordinated activity in the upper and lower airway muscles of the fetal lamb in utero. Pediatr Res. 1988 Mar;23(3):257-61. doi: 10.1203/00006450-198803000-00005. PMID 3353170
- [Derived] Ozkan D, Gonen E, Akkaya T, Bakir M. Popliteal block for lower limb surgery in children with cerebral palsy: effect on sevoflurane consumption and postoperative pain (a randomized, double-blinded, controlled trial). J Anesth. 2017 Jun;31(3):358-364. doi: 10.1007/s00540-017-2318-2. Epub 2017 Feb 14. PMID 28197774